CLINICAL TRIAL: NCT02669589
Title: Regional Citrate Versus Systemic Heparin Anticoagulation for Continuous Renal Replacement Therapy in Critically Ill Patients With Acute Kidney Injury
Brief Title: Investigating Different Anticoagulants for Renal Replacement Therapy
Acronym: RICH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: University of Leipzig (Other); German Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKM 14_0066; 2014-004854-33 (EudraCT Number); 03-AnIt-14 (Other: Dept. of Anesthesiology, Intensive Care and Pain Medicine)
Record Dates: First submitted 2016-01-19; First posted 2016-02-01 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2019-02

CONDITIONS: Acute Kidney Injury
Keywords: CRRT; AKI; anticoagulation; KDIGO
MeSH Terms: conditions — Acute Kidney Injury | interventions — Heparin; Citric Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- heparin anticoagulation (Active Comparator): Systemic anticoagulation of the continuous renal replacement therapy with heparin.
  Dose will be titrated to maintain aPTT (activated partial thromboplastin time) between 45-60s)
  Interventions: Drug: Heparin
- citrate anticoagulation (Experimental): Regional anticoagulation of the continuous renal replacement therapy with citrate.
  Target posthemofilter ionized calcium level: 0.25-0.35 mmol/l
  Interventions: Drug: Citrate

INTERVENTIONS:
Drug: Heparin
  Arms: heparin anticoagulation
Drug: Citrate
  Arms: citrate anticoagulation

SUMMARY:
The aim of this study is to evaluate the effect of regional citrate anticoagulation within the scope of continuous renal replacement (CRRT) in critically ill patients with acute kidney injury (AKI) on filter life span and 90-day all cause mortality.

DETAILED DESCRIPTION:
Purpose of clinical trial:

To evaluate the effect of regional citrate anticoagulation within the scope of continuous renal replacement (CRRT) in critically ill patients with acute kidney injury (AKI) on filter life span and 90-day all cause mortality.

Patient population: critically ill patients with acute kidney injury requiring renal replacement therapy.

Primary objective:

Anticoagulation of the extracorporeal circuit is required in continuous RRT (CRRT). To this date, it is not clear which anticoagulant should be used for CRRT. Regional citrate anticoagulation (RCA) for CRRT in critically ill patients with AKI prolongs filter life span and reduces 90-day all cause mortality by approximately 8% (from 48% to 40%) compared to systemic heparin anticoagulation for CRRT

ELIGIBILITY:
Inclusion Criteria:

1. Critically ill patients with clinical indication for CRRT (clinical decision to use continuous RRT due to hemodynamic instability)

   Or

   Severe acute kidney injury (KDIGO 3-classification) despite optimal resuscitation
2. At least one of the following conditions

   * Sepsis or septic shock
   * Use of catecholamines (norepinephrine or epinephrine ≥ 0.1 µg/kg/min or norepinephrine ≥ 0.05 µg/kg/min + dobutamine (any dose) or norepinephrine ≥ 0.05 µg/kg/min + vasopressin (any dose) or epinephrine ≥ 0.05 µg/kg/min + norepinephrine ≥ 0.05 µg/kg/min)
   * Refractory fluid overload: worsening pulmonary edema: PaO2/FiO2 < 300 mmHg and/or fluid balance > 10% of body weight)
3. 18-90 years old
4. Intention to provide full intensive care treatment for at least 3 days
5. Written informed consent of the patient or the legal representatives or the authorized representative or the inclusion due to an emergency situation

Exclusion Criteria:

1. Patients with increased bleeding risk (e.g. an active bleeding from ulcers in the gastro-intestinal tract, hypertension with a diastolic blood pressure higher than 105 mm Hg, injuries (intracranial hemorrhage, aneurysm of brain arteries) of or surgical procedures on the central nervous system if a heparinization with a target aPTT 45-60 s is not allowed by the treating neurologist or neurosurgeon, severe retinopathies, bleeding into the vitreum, ophthalmic surgical procedures)) or injuries, active tuberculosis; infective endocarditis)
2. Disease or organ damage related with hemorrhagic diathesis (coagulopathy, thrombocytopenia, severe liver or pancreas disease)
3. Dialysis-dependent chronic kidney insufficiency
4. Need of therapeutic systemic anticoagulation
5. Allergic reaction to one of the anticoagulants or ingredients, Heparin-induced thrombocytopenia
6. AKI caused by permanent occlusion or surgical lesion of the renal artery
7. AKI caused by (glomerulo)nephritis, interstitial nephritis, vasculitis or postrenal obstruction
8. Do-not-resuscitate order
9. Hemolytic-uremic syndrome/thrombotic thrombocytopenic purpura
10. Persistent and severe lactate acidosis in the context of an acute liver failure and/or shock
11. Kidney transplant within the last 12 months
12. Pregnancy and nursing period
13. Abortus imminens
14. No hemofiltration machine free for use at the moment of inclusion
15. Participation in another clinical intervention trial in the last 3 months
16. Persons with any kind of dependency on the investigator or employed by the sponsor or investigator
17. Persons held in an institution by legal or official order

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 638 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
CRRT-filter life span in hours | during continuous renal replacement therapy up to 1 year
  It will be reported how long the filter will be used during CRRT
Overall survival in a 90day follow-up period | 90 days

SECONDARY OUTCOMES:
ICU length of stay in days | up to 1 year
  The primary ICU stay will be documented.
Hospital length of stay in days | up to 1 year
duration of renal replacement therapy | 1 year
  within 1 year after randomization
Bleeding complication | intraoperative
Number of patients with administration of red blood cells | intraoperative
Rate of infection | during primary ICU stay up to 1 year
Major adverse kidney events | day 28, 60, 90 and after 1 year after start of CRRT
Complications of therapy | intraoperative
Recovery of renal function | day 28, 60, 90 and 1 year after start of CRRT
  The recovery of renal function will be defined as composite endpoint consisting of lack of dialysis dependency and serum creatinine level no more than 0.5 mg/dl above the baseline value)
Number of participants with hemodialysis | day 28, 60, 90 and 1 year after start of CRRT
Mortality | day 28, 60 and 1-year

OTHER OUTCOMES:
SOFA Scores (Sepsis-related Organ Failure Assessment score) | day 1-14, 21 and 28 during ICU stay
serum creatinine level in mg/dL | Day 0, day 1, day 3, day 5 and 1 day after CRRT cessation
plasma urea concentration in mg/dl | Day 0, day 1, day 3, day 5 and 1 day after CRRT cessation
glomerular filtration rate | Day 0, day 1, day 3, day 5 and 1 day after CRRT cessation

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Zarbock, MD, Study Chair — University Hospital Muenster
Locations (31):
- Germany (31):
  - University Hospital Aachen, Aachen
  - Klinikum Augsburg, Augsburg
  - HELIOS Klinikum Bad Saarow, Dept. of Intensive Care, Bad Saarow
  - Charité Berlin, Dept. of Anesthesiology and Intensive Care Medicine, Berlin
  - Charité Berlin CCM, Medical Department, Division of Nephrology, Berlin
  - Charité Berlin CCV, Medical Department, Division of Nephrology, Berlin
  - Evangelisches Klinikum Bethel gGmbH, Bielefeld
  - Universitätsklinikum Knappschaftskrankenhaus Bochum, Bochum
  - University Hospital Bonn, Dept.of Anesthesiology and Intensive Care Medicine, Bonn
  - Klinikum Köln-Merheim, Medizinische Klinik I, Cologne
  - University Hospital Duesseldorf, Dept. of Anaesthesiology, Düsseldorf
  - University Hospital Düsseldorf, Dept. of Nephrology, Düsseldorf
  - University Hospital Erlangen, Erlangen
  - University Hospital Essen, Dept. for Nephrology, Essen
  - University Hospital Frankfurt, Dept. of Anesthesiology, Intensive-Care Medicine and Pain Therapy, Frankfurt
  - University Hospital Gießen, Dept. of Anesthesiology and Intensive Care, Giessen
  - University Medical Center Göttingen, Dept. for Anesthesiology, Göttingen
  - University Medicine Greifswald, Greifswald
  - University Hospital Halle, Dept. of Anesthesiology and Intensive Care, Halle
  - University Medical Center Hamburg-Eppendorf, Dept. of Intensive Care, Hamburg
  - University Hospital Heidelberg, Dept. of Anesthesiology, Heidelberg
  - University Hospital Jena, Dept. of Anesthesiology and Intensive Care Medicine, Jena
  - University Hospital Schleswig-Holstein, Campus Kiel, Dept. for Anaesthesiology and Intensive Care, Kiel
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsmedizin Mainz, Mainz
  - Technical University of Munich University Hospital, Dept. for Anaesthesiology, München
  - University Hospital Muenster, Münster
  - Klinikum Nürnberg, Nuremberg
  - University Hospital Regensburg, Dept. of Surgery, Regensburg
  - Municipal Hospital Solingen, Dept. for Nephrology and General Internal Medicine, Solingen
  - University Hospital Tuebingen, Tübingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] von Groote T, Albert F, Meersch M, Koch R, Gerss J, Arlt B, Sadjadi M, Porschen C, Pickkers P, Zarbock A; RICH investigators. Evaluation of Proenkephalin A 119-159 for liberation from renal replacement therapy: an external, multicenter pilot study in critically ill patients with acute kidney injury. Crit Care. 2023 Jul 10;27(1):276. doi: 10.1186/s13054-023-04556-w. PMID 37430375
- [Derived] Tsujimoto H, Tsujimoto Y, Nakata Y, Fujii T, Takahashi S, Akazawa M, Kataoka Y. Pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2020 Dec 14;12(12):CD012467. doi: 10.1002/14651858.CD012467.pub3. PMID 33314078
- [Derived] Zarbock A, Kullmar M, Kindgen-Milles D, Wempe C, Gerss J, Brandenburger T, Dimski T, Tyczynski B, Jahn M, Mulling N, Mehrlander M, Rosenberger P, Marx G, Simon TP, Jaschinski U, Deetjen P, Putensen C, Schewe JC, Kluge S, Jarczak D, Slowinski T, Bodenstein M, Meybohm P, Wirtz S, Moerer O, Kortgen A, Simon P, Bagshaw SM, Kellum JA, Meersch M; RICH Investigators and the Sepnet Trial Group. Effect of Regional Citrate Anticoagulation vs Systemic Heparin Anticoagulation During Continuous Kidney Replacement Therapy on Dialysis Filter Life Span and Mortality Among Critically Ill Patients With Acute Kidney Injury: A Randomized Clinical Trial. JAMA. 2020 Oct 27;324(16):1629-1639. doi: 10.1001/jama.2020.18618. PMID 33095849
- [Derived] Meersch M, Kullmar M, Wempe C, Kindgen-Milles D, Kluge S, Slowinski T, Marx G, Gerss J, Zarbock A; SepNet Critical Care Trials Group. Regional citrate versus systemic heparin anticoagulation for continuous renal replacement therapy in critically ill patients with acute kidney injury (RICH) trial: study protocol for a multicentre, randomised controlled trial. BMJ Open. 2019 Jan 21;9(1):e024411. doi: 10.1136/bmjopen-2018-024411. PMID 30670518